CLINICAL TRIAL: NCT05052710
Title: A Fixed Sequence, Open-label Study to Assess the Effect of Multiple Doses of AZD4831 on the Pharmacokinetics of Oral Midazolam (a CYP450 3A Probe) in Healthy Subjects
Brief Title: Study to Assess the Effect of AZD4831 on the Pharmacokinetics (Drug Behavior in the Body) of Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6580C00012
Record Dates: First submitted 2021-09-14; First posted 2021-09-22 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteers
Keywords: Cardiovascular Disease; Drug-drug interaction; Pharmacokinetics; Myeloperoxidase inhibitor; Fixed-sequence
MeSH Terms: conditions — Cardiovascular Diseases | interventions — AZD4831; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Subjects will receive midazolam on Day 1 and AZD4831 once daily from Days 2 to 10, and AZD4831 plus midazolam on Day 11.
  Interventions: Drug: AZD4831; Drug: Midazolam

INTERVENTIONS:
Drug: AZD4831 — Subjects will receive oral doses once daily from Days 2-11.
Drug: Midazolam — Subjects will receive oral single doses on Day 1 and Day 11.

SUMMARY:
The study is an open-label, fixed-sequence, cross-over study conducted at a single Clinical Unit to assess the pharmacokinetics (PK) of midazolam in healthy male and female (non-childbearing potential) subjects when administered alone and in combination with AZD4831 after multiple doses (once daily) of AZD4831 for 10 consecutive days.

DETAILED DESCRIPTION:
The study will consist of 2 treatment periods and will comprise:

* A Screening period of maximum 28 days;
* Treatment Period 1 and Treatment Period 2:

Treatment Period 1: Midazolam only (Day 1). Treatment Period 2: AZD4831 only (Days 2 to 10, once daily dosing) and AZD4831 plus midazolam (Day 11).

- A final Follow-up Visit after the last administration of investigational medicinal product (IMP) (Day 20 [± 1 day]).

Each subject will be involved in the study for approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects with suitable veins for cannulation or repeated venepuncture.
* Males must be willing to use appropriate contraception methods.
* Females must not be lactating and must be of non-childbearing potential, confirmed at Screening.
* Have a body mass index between 18.5 and 30 kg/m^2 (inclusive) and weigh at least 50 kg and no more than 100 kg (inclusive) at Screening.

Exclusion Criteria:

* History of any clinically significant disease or disorder.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* A positive Corona Virus Disease 2019 test at Screening or admission to the Clinical Unit on Day -1.
* Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results.
* Any clinically significant abnormal findings in vital signs.
* clinically significant abnormalities on 12-lead electrocardiogram.
* Any positive result at the Screening Visit for Hepatitis B surface antigen, hepatitis C virus antibody, and human immunodeficiency virus antibody.
* Known or suspected history of drug abuse in the last 2 years.
* Current smokers or those who have smoked or used nicotine products within the 3 months prior to the Screening Visit.
* Known or suspected history of alcohol or drug abuse.
* Use of any prescribed or non-prescribed medication.
* Subjects with acute pulmonary insufficiency, marked neuromuscular respiratory weakness, obsessional states, phobic states, sleep apnoea syndrome, or unstable myasthenia gravis.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigatoror history of hypersensitivity to drugs with a similar chemical structure or class to AZD4831 or midazolam.
* History or ongoing allergy/hypersensitivity to drugs(including but not limited to rash, angioedema, acute urticaria).
* Subjects who, in the opinion of the Investigator, have any clinically significant skin condition.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration time curve from zero to infinity (AUCinf) of Midazolam | Days 1, 2, 11, and 12
  Effect of AZD4831 on AUCinf of Midazolam will be assessed.
Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) of Midazolam | Days 1, 2, 11, and 12
  Effect of AZD4831 on AUClast of Midazolam will be assessed.
Maximum observed plasma (peak) drug concentration (Cmax) of Midazolam | Days 1, 2, 11, and 12
  Effect of AZD4831 on Cmax of Midazolam will be assessed.

SECONDARY OUTCOMES:
Time to reach peak or maximum observed concentration or response following drug administration (tmax) of Midazolam and AZD4831 | Midazolam:Days 1, 2, 11, and 12; AZD4831:Days 2-12
  tmax of Midazolam and AZD4831 will be assessed.
Half life associated with terminal slope (λz) of a semi logarithmic concentration timecurve (t½λz) of Midazolam and AZD4831 | Midazolam:Days 1, 2, 11, and 12; AZD4831:Days 2-12
  t½λz of Midazolam and AZD4831 will be assessed.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) of Midazolam and AZD4831 | Midazolam:Days 1, 2, 11, and 12; AZD4831:Days 2-12
  CL/F of Midazolam and AZD4831 will be assessed.
Apparent volume of distribution based on terminal phase (Vz/F) of Midazolam | Days 1, 2, 11, and 12
  Vz/F of Midazolam will be assessed.
Area under the plasma concentration-curve across the dosing interval (AUCtau) of AZD4831 | Days 2-12
  AUCtau of AZD4831 will be assessed.
Cmax of AZD4831 | Days 2-12
  Cmax of AZD4831 will be assessed.
Daily pre-dose plasma concentration (CpreD3 up to CpreD10) of AZD4831 | Days 3-10
  Pre-dose plasma concentration of AZD4831 will be assessed.
Plasma concentration 24 hours post the Day 10 dose (C24h) of AZD4831 | Day 11
  Plasma concentration of AZD4831 will be assessed.
Number of patients with adverse events (AE) and serious AEs (SAE) | From Screening (Day -28 to Day -2) until Follow-up Visit (Day 20)
  Safety and tolerability of AZD4831 alone and in combination with midazolam will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home